CLINICAL TRIAL: NCT03083002
Title: Study of Hepatocellular Carcinoma Risk in Patient With Liver Cirrhosis
Brief Title: Risk of Hepatocellular Carcinoma in Patient With Liver Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, ERICA VILLA, Professor, University of Modena and Reggio Emilia
Other Study IDs: UNIRER 2
Record Dates: First submitted 2017-03-07; First posted 2017-03-17 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-03

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Purpose of the study is to determine transcriptomics, metabolomics and proteomics features of liver cirrhotic tissue in patients with hepatocellular carcinoma (HCC) and to find a correlation with the risk of developing HCC and survival.

DETAILED DESCRIPTION:
Patients will be enrolled after hepatic ultrasonography control and they will be submitted to hepatic vein pressure gradient and liver biopsy.

The study have four research lines:

Task # 1: transcriptomic characterization of liver tissue. During hepatic vein pressure gradient , liver tissue will be extracted with transjugular catheter equipped with a biopsy device. Tissue will be used to extract microRNA to define molecular signature.

Task # 2: Proteomic characterization of liver tissue. Protein expression changes will be analyze with MALDI-TOF

Task # 3: Metabolomic features on serum of patient with cirrhosis. Metabolomics is defined as the quantitative measurement of the dynamic multiparametric response of living systems to pathophysiological stimulus or genetic modification. Principal objective of this activity will be identify metabolites deregulated with metabolomic approach and clarify any new pathways involved in the evolution of cirrhosis to hepatocellular carcinoma.

The metabolomic analysis will be performed on sera collected in patients with cirrhosis at baseline.

Task # 4: Transcriptomic characteristics of newly diagnosed HCC. New diagnosis of hepatocellular carcinoma will undergo an eco-assisted liver biopsy. A tissue sample will be dedicated to the extraction of 'RNA. Patients will then undergo elective treatment according to international guidelines. The course of the disease and the results of therapeutic interventions will be recorded and correlated with the molecular data. Molecular signature will be obtain.

ELIGIBILITY:
Inclusion Criteria:

* Obtaining written informed consent
* Liver cirrhosis
* Aged between 18 and 75 years
* Absence of exclusion criteria

Exclusion Criteria:

* HCC
* HIV
* Pregnancy
* Portal vein thrombosis
* Liver Transplant
* Patients' refusal to participate in clinical research

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver cirrhosis will be selected. After obtaining informed consent they will be submitted to hepatic biopsy,blood sample, HVPG with combined right heart catheterization and every 6 months to ultrasound.
  Patients will be followed for 24 months thereafter or until the diagnosis of HCC, whichever comes first. In case of onset of HCC, will be performed a eco-guided biopsy.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2013-05; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Transcriptomics characterization of liver tissue: the purpose is molecular evaluation of possible predisposing factors to development of hepatocellular carcinoma in patients with cirrhosis. | December 2017
  RNA sample will be collected from patients and used to obtained transcriptomic profile through microarray and microRNA. Patients will be submitted to hepatic vein pressure gradient and combined right heart catheterization. During this standard procedure liver tissue will be taken and treated for extraction of RNA.
  In order to obtain microarray RNA extracted will be analyzed with single color hybridization of human RNA on Agilent Whole Human Genome Oligo whereas, the extraction of microRNA will be made starting from RNA extracted with mirVana miRNA Isolation kit.

SECONDARY OUTCOMES:
Proteomic characterization of liver tissue: the objective is to understand if there is a relationship between emergence of HCC and alterations of protein expression in cirrhotic liver. | DECEMBER 2017
  Modifications of protein expression will be examined by two-dimensional electrophoresis and MALDI-TOF.
Metabolomic features of patient with cirrhosis: principal aim of this task is to identify particular metabolites and potential new pathway involved in the evolution of cirrhosis to hepatocellular carcinoma | DECEMBER 2017
  Analysis will be conducted on sera collected during the screening. These samples will be examined using liquid chromatography and mass spectrometry in order to obtain the identification of main components and their mass than, the informations will be analyzed by MarkerLynxTM software
Transcriptomics characteristics of newly diagnosed hepatocellular carcinoma: the purpose is to verify if we can predict the survival of patients considering the molecular features of HCC at first diagnosis. | DECEMBER 2017
  Patients with new diagnosis of hepatocellular carcinoma will be subjected to liver biopsy. A part of biopsy will be used to extract RNA and we will try to identify molecular signature through qRT / PCR (polymerase chain reaction) and using a set of 12 up- regulated and 10 down - regulated genes previously identified.

CONTACTS AND LOCATIONS:
Overall Officials: ERICA VILLA, Principal Investigator — Università di Modena e Reggio Emilia
Locations (1):
- Azienda Ospedaliera Universitaria Policlinico Di Modena, Modena, MO, Italy

IPD SHARING:
Plan to Share IPD: No